CLINICAL TRIAL: NCT03611764
Title: The Mindfulness Pilot Project: The Effects of a Body Scan Activity on Bone Marrow Transplant Patients and Their Caregivers
Brief Title: Body Scan Activity on Bone Marrow Transplant Patients and Their Caregivers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Only 5 caregivers decided to participate
Sponsor: Washington University School of Medicine (Other)
Collaborators: Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 201803060
Record Dates: First submitted 2018-07-19; First posted 2018-08-02 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Hematological Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Whole Body Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1: Body Scan (Experimental): * The mindfulness-based intervention (MBI) of the Body Scan is expected to take 20 minutes
  * Participants will then be guided through the Body Scan. Beginning with awareness of sensations of the left toe, patients will be asked to observe these sensations without judgment, simply noticing and allowing them. Awareness of sensations will continue up through the left leg, then from the right toe up the right leg, then abdomen and chest, then fingertips to arms, then neck, and finally the head. After completing the Body Scan, participants will be given several minutes of quiet to reflect upon how they feel. After opening their eyes, participants will be given the opportunity to discuss and ask questions.
  * Caregivers will be encouraged to practice with the patient or on their own, in an additional space on the floor called the Zen Den
  Interventions: Behavioral: Body Scan; Other: Rotterdam Symptom Checklist; Other: Practice Logs

INTERVENTIONS:
Behavioral: Body Scan — -All efforts will be made to normalize their experience: for example, the desire to open their eyes, thinking about other things, wanting to move around - these are all normal and participants will be encouraged to become interested in and curious about, and to allow these natural tendencies
Other: Rotterdam Symptom Checklist — * 39 Likert-scale items, including physical and psychological symptoms (30 questions), daily function (8 questions), and overall valuation of life (one question)
  * For the 30 questions pertaining to symptoms, the four-item Likert scale ranges from 'not at all=1' to 'very much=4'; the higher the total score, the greater the score, the higher the level of distress. The single question pertaining to overall valuation of life asks participants to circle one of the seven items, ranked from "extremely poor" to "excellent"
  Other Names: RSCL
Other: Practice Logs — -Describe frequency of the Zen Den

SUMMARY:
This study will address whether teaching the Body Scan exercise to cancer patients with hematological malignancies and their caregivers during an inpatient hospitalization improves reported physical and psychological symptoms after a two-week period. Giving patients and caregivers the opportunity to learn mindfulness and the tools to practice on their own is expected to lead to a decrease in stress and anxiety, and help empower patients and caregivers to better cope with stress in the future.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary & self-selected patients and caregivers
* Located on the leukemia/lymphoma/bone marrow transplant floor at Barnes Jewish Hospital

Exclusion Criteria:

-Patients requiring a language translator or interpreter will be excluded from the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Measure of distress in patients measured by the RSCL scores | Through 2 weeks
  -Inferential statistics will be used to analyze the Rotterdam Symptom Checklist (RSCL)
Measure of distress in caregivers measured by the RSCL scores | Through 2 weeks
  -Inferential statistics will be used to analyze the Rotterdam Symptom Checklist (RSCL)

SECONDARY OUTCOMES:
Frequency of body scan practice | Through 2 weeks
  -Practice Logs will be used to notate frequency of body scan practice

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Compernolle, BSN, RN, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu